CLINICAL TRIAL: NCT00855049
Title: A Randomized Crossover Study to Determine the Pharmacokinetics of Intranasally Administered Acetaminophen in Healthy Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain FDA approval
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry); American College of Medical Toxicology (Other)
Responsible Party: Sing-Yi Feng, MD, University of Texas Southwestern Medical Center/Children's Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 052008-076
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics; Acetaminophen; Intranasal; Absorption
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intranasal acetaminophen administration
  Interventions: Drug: Acetaminophen
- 2 (Active Comparator): Oral acetaminophen administration
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Intranasal acetaminophen administration
  Other Names: Tylenol; Paracetamol
  Arms: 1
Drug: Acetaminophen — Oral acetaminophen administration
  Other Names: Tylenol; Paracetamol
  Arms: 2

SUMMARY:
This study is being done to determine the systemic absorption of nasally inhaled acetaminophen (Tylenol®) versus orally ingested acetaminophen by comparing the serum drug concentrations of the two groups obtained at various times after study drug administration.

DETAILED DESCRIPTION:
This study is aimed at addressing a significant void in the current literature regarding nasally administered acetaminophen pharmacokinetics. The pharmacokinetics of acetaminophen following oral and rectal administration have been well studied but to date there are no published studies determining the pharmacokinetics of acetaminophen following intranasal administration. This route is currently popular among heroin users. Understanding the pharmacokinetics of nasally administered acetaminophen will help physicians address the important clinical implications of acetaminophen toxicity in this population.

Ten healthy adult volunteers age 18 to 45 years will be recruited for this pilot project. Study participants will be randomized in permuted blocks to receive either oral or intranasal administration of a standardized 500 mg dose of acetaminophen. Blood samples will be drawn from a peripheral intravenous catheter at 0, 5, 15, 30, 45, 60, 90, 120, 150, 240, 360, and 480 minutes after study drug administration and sent to the laboratory for determination of serum acetaminophen concentration. After a one week washout period, each participant will cross over to receive 500 mg of acetaminophen via the remaining route of administration in the second arm of the study. The serial acetaminophen concentrations will be utilized to perform pharmacokinetic calculations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18 to 45 years of age

Exclusion Criteria:

* Known hypersensitivity to acetaminophen
* Prior dosing of acetaminophen or product containing acetaminophen in the preceding 7 days
* Hepatic insufficiency and/or failure, or any known liver disease
* History of nasal polyps
* History of nasal trauma in past 14 days
* History of nasal bleeding in past 14 days
* History of asthma, emphysema or any serious respiratory diseases
* Pregnancy or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Serum acetaminophen levels | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sing-Yi Feng, MD, Principal Investigator — UT Southwestern/Children's Medical Center
Locations (1):
- UT Southwestern, Dallas, Texas, United States